CLINICAL TRIAL: NCT07379905
Title: A Randomized Trial of MODUCARE Versus Wait-and-See Approach for Histologically Proven Low-grade Cervical Intraepithelial Neoplasia (CIN1)
Brief Title: MODUCARE Versus Wait-and-See Approach for Histologically Proven Low-grade Cervical Intraepithelial Neoplasia (CIN1)
Acronym: MODUCIN1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: INPA S.A. (Unknown)
Responsible Party: Principal Investigator, Dimitrios Zouzoulas, Gynecological Oncologist, MSc, PhD, FEBS-BS, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-Β2015-518
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Low-grade Cervical Intraepithelial Neoplasia; Moducare

STUDY DESIGN:
Intervention Model Description: * ARM A: Control Arm for Wait-and-See approach
  * ARM B: Intervation Arm for MODUCARE oral capsules, dosage 2 x 3 for 1 month and 1 x 3 for 5 months (total 6 months, as per instructions provided by the manufacturer)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: Control Arm (No Intervention): Wait-and-See approach
- ARM B: Intervention Arm (Experimental): MODUCARE oral capsules., dosage 2 x 3 for 1 month and 1 x 3 for 5 months (total 6 months, as per instructions provided by the manufacturer)
  Interventions: Dietary Supplement: MODUCARE

INTERVENTIONS:
Dietary Supplement: MODUCARE — MODUCARE is classified as a natural dietary supplement, specifically an immune support supplement containing a patented blend of plant sterols and sterolins, primarily beta-sitosterol and beta-sitosterol glucoside, derived from plant sources.
  Arms: ARM B: Intervention Arm

SUMMARY:
MODUCIN-1 (MODUcare for CIN1) is a prospective, single center, open-label, randomized trial that its purpose is to compare MODUCARE versus Wait-and-See Approach for the regression rate of histologically proven low-grade Cervical Intraepithelial Neoplasia (CIN1).

DETAILED DESCRIPTION:
Human Papillomavirus (HPV) is causally associated with cervical cancer and precancerous lesions (dysplasias) of the cervix. These lesions are detected mainly in the transformation zone and are diagnosed with colposcopy and biopsy confirmation. In high-grade lesions conization (surgical removal of a cone tissue form the cervix) is the therapy of choice, but in low-grade lesions monitoring and no-treatment is preferred. However, this wait-and-see approach can be assisted by pharmaceutical treatment, like MODUCARE.

MODUCARE is classified as a natural dietary supplement, specifically an immune support supplement containing a patented blend of plant sterols and sterolins, primarily beta-sitosterol and beta-sitosterol glucoside, derived from plant sources. It is taken orally, 2 capsules three times daily for the first month and then 1 capsule three times daily for next 5 months (in total 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CIN1
* Any HPV status (negative, positive: high or low risk)
* Any Pap test result
* Age 18 - 85 years old
* ECOG Performance status 0 - 1

Exclusion Criteria:

* Pregnancy
* Low likelihood of patient compliance to treatment protocol and follow-up
* Previous operation to the cervix
* Previous pelvic malignancy
* Pre-existing histologically proven CIN1 > 12 months
* Pre-existing histologically proven CIN2 and/or CIN3
* Hypersensitivity to trial medication

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 182 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Regression rate of CIN1 | 6 months after randomization

SECONDARY OUTCOMES:
Regression rate of CIN1 | 12 months after randomization
Progression rate of CIN1 | 6 & 12 months after randomization
Treatment related adverse events | : 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Tsolakidis, Dr.Prof., Principal Investigator — Aristotle University Of Thessaloniki

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD only after contact with the principal investigator for the synthesis of future studies.